CLINICAL TRIAL: NCT05816109
Title: The Effect of Superficial Cervical Plexus Block on Postoperative Recovery Quality and Pain in Anterior Cervical Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, associate professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022/09
Record Dates: First submitted 2023-01-19; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain
Keywords: Recovery Quality; Postoperative Pain; Superficial cervical block; Cervical block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial cervical block (Experimental): Superficial Cervical Block
  Interventions: Diagnostic Test: superficial cervical block
- without superficial cervical block (Active Comparator): Without superficial cervical block
  Interventions: Diagnostic Test: without superficial cervical block

INTERVENTIONS:
Diagnostic Test: superficial cervical block — After anesthesia and surgical procedures, bilateral superficial cervical plexus block will be applied to the lower border of the sternocleidomastoid muscle, accompanied by ultrasonography. After cleaning the area with povidone iodine before the block, the sternocleidomastoid muscle and carotid artery and other vascular structures are determined using a linear ultrasound probe. Local anesthetic will be administered between the lower border of the sternocleidomastoid muscle and the upper border of the prevertebral fascia with the help of an insulated needle designed for peripheral block procedures. The location of the needle will be confirmed by hydrodissection method with saline before local anesthesia is given. After the location of the needle is confirmed, 2 ml of saline will be injected, followed by 10 ml of 0.5% bupivacaine. The deep cervical fascia of the superficial lamina will appear to open.
  Arms: Superficial cervical block
Diagnostic Test: without superficial cervical block — patients who underwent anterior cervical surgery and did not undergo superficial cervical block
  Arms: without superficial cervical block

SUMMARY:
The Effect of Superficial Cervical Plexus Block on Postoperative Recovery Quality and Pain in Anterior Cervical Spinal Surgery

DETAILED DESCRIPTION:
The study was designed as a double-blind, prospective randomized controlled trial.

Blindness; The healthcare professionals who will monitor the patient's pain in the post-operative period will not know whether the superficial cervical plexus block is applied to the patients. Randomization of the patients was planned using computer aided. It is envisaged that 20 participants will be included in the patient group that will have a superficial cervical plexus block and will not have a superficial cervical plexus block. The current pain status in the postoperative period in the patient groups that will or will not have a superficial cervical plexus block is determined by NRS (Numerical rating scale) at rest and in motion at certain hour intervals ( 30.min,1.,6.,12.,24. hours) will be done, when the patients' NRS scores are 4 and above, an additional intravenous analgesic will be administered, and the number of bolus doses with PCA in the first 24 hours will be recorded. The quality of recovery (QoR-40) scoring system will be evaluated at the postoperative 24th hour of both patients with and without superficial cervical plexus block. In addition, the hemodynamic values of the patients will be recorded in these intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar spinal surgery under elective conditions
* ASA I-III
* Between 18-75 ages

Exclusion Criteria:

refuse during registration

* request to be dismissed from study
* failure to give informed consent
* emergency surgery
* bleeding diathesis
* Presence of contraindications to the LA agents used in this study chronic use of opioids psychiatric disorders the presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Qor-40 test (The recovery quality test) | 24 th hour
  For this purpose, patients will be subjected to the Short Form-40- test , which is a short scale of postoperative recovery quality at first 24th hour. Minimum score is 40=bad, maximum score is 200=good

SECONDARY OUTCOMES:
NRS (Numerical rating scale) | 30 minutes,1st hour,6th hour,12th hour and 24th hour]
  It is pain intensity determination system based on the system where the person tells a point between 0=(no pain), 10= (unbearable pain) and to describe their pain.
Postoperative pain | 30 minutes, 1st hour, 6th hour, 12th hourand 24th hour
  Postoperative opioid consumotions on the pca (patient controlled analgesia) device of the patients will be recorded in Postoperative 30. min, 1., 6., 12., 24. Opioid consumptions on the pca device of the patients will be recorded in 30. min, 1., 6., 12., 24. hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Faculty of Medicine, Aydin, Turkey (Türkiye)